CLINICAL TRIAL: NCT04550559
Title: Evaluation of the Effect of Masturbation on Distal Ureteral Stones: A Prospective Randomized Controlled Study
Brief Title: Rate of Spontaneous Stone Passage as Assessed Using Urinary Ultrasonography and Direct Urinary System Radiography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Avrasya University (Other)
Responsible Party: Principal Investigator, Hasan Turgut, urolog dr ,Principal Investigator, Avrasya University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: masturbation and stone
Record Dates: First submitted 2020-09-01; First posted 2020-09-16 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Ureteral Calculi; Masturbation
MeSH Terms: conditions — Ureteral Calculi; Masturbation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Active Comparator): The patients in group 1 were instructed to masturbate at least 3-4 times a week
  Interventions: Procedure: Endoscopic ureterolitotripsy
- Group 2 (Other): The patients in group 2 were prescribed oral tamsulosin 0.4 mg once daily
  Interventions: Procedure: Endoscopic ureterolitotripsy
- Group 3 (No Intervention): The patients in group 3 acted as controls and received only standard medical therapy

INTERVENTIONS:
Procedure: Endoscopic ureterolitotripsy — Endoscopic ureterolithotripsy
  Arms: Group 1; Group 2

SUMMARY:
To evaluate the effect of masturbation on the spontaneous expulsion of distal ureteral stones 5-10 mm in size.

DETAILED DESCRIPTION:
This prospective randomized controlled study was performed between February 2018 and March 2020 after obtaining ethics committee approval.A total of 128 men with distal ureteral stones were randomly divided into 3 groups. All patients received standard medical therapy. Patients in group 1 (n=43) were instructed to masturbate at least 3-4 times a week, patients in group 2 (n=41) received tamsulosin 0.4 mg/day, and patients in group 3 (controls, n=44) received standard medical therapy alone. Rates of expulsion, need for analgesic, and ureterorenoscopic lithotripsy were compared between the groups.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years
* presenting with renal colic and inguinal or lumbar pain
* being diagnosed as having distal ureteral stones ≥5 mm and <10 mm in size

Exclusion Criteria:

* age <18 years,
* stones <5 mm or ≥10 mm in size,
* intermediate (stones on the ureter-iliac artery cross)
* proximal ureteral stones, multiple ureteral stones,
* presence of urinary infection,
* renal insufficiency,
* high creatinine level,
* severe hydroureteronephrosis,
* history of open or endoscopic ureteral surgery,
* vesicoureteral reflux,
* neurogenic bladder,
* erectile dysfunction,
* inability or refusal to masturbate for any reason (such as religious beliefs)

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
The rates of spontaneous distal ureteral stone (5-10 mm size) passage after 4 weeks masturbation | 4 weeks
  The rates of spontaneous distal ureteral stone (5-10 mm size) passage of patients who were instructed to masturbate at least 3-4 times a week (Group1); received tamsulosin 0.4 mg/day (Group2); received standard medical therapy alone Group3.

CONTACTS AND LOCATIONS:
Overall Officials: Hasan Turgut, Dr, Principal Investigator — Avrasya University Health Science Faculty
Locations (1):
- Hasan Turgut, Trabzon, Turkey (Türkiye)